CLINICAL TRIAL: NCT00944528
Title: Single Dose Partial Breast Radiotherapy Using Extra-cranial Radiosurgery in Patients With Early Stage Breast Cancer - a Phase I Dose Escalation Study
Brief Title: Single Dose Partial Breast Radiotherapy
Acronym: RSU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00015617
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: Cancer of Breast; Cancer of the Breast; Neoplasms, Breast; Single dose radiation; Radiotherapy; Preoperative
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single dose radiosurgery: Dose Level 1 (Experimental): A single 15 Gy dose of radiation given in radiosurgery technique about 10 days before lumpectomy.
  Interventions: Radiation: Radiosurgery
- Single dose radiosurgery: Dose Level 2 (Experimental): A single 18 Gy dose of radiation given in radiosurgery technique about 10 days before lumpectomy.
  Interventions: Radiation: Radiosurgery
- Single dose radiosurgery: Dose Level 3 (Experimental): A single 21 Gy dose of radiation given in radiosurgery technique about 10 days before lumpectomy.
  Interventions: Radiation: Radiosurgery

INTERVENTIONS:
Radiation: Radiosurgery — Single dose or radiation in 15Gy, 18Gy or 21Gy
  Other Names: External beam radiation therapy

SUMMARY:
This study seeks to determine the maximum tolerated dose of a single-dose partial breast radiation given before lumpectomy using a radiosurgery technique. Lumpectomy will be performed within 3 weeks (+/- 1 week) of completing radiation.

DETAILED DESCRIPTION:
This study will assess the safety of partial breast radiosurgery as measured by the incidence of acute toxicity and wound healing complications in three dose cohorts.

Patients will be enrolled in cohorts of 8 patients starting at dose level 1 (15 Gy). If 2 or more dose limiting toxicities (DLTs) are observed at dose level 1, the trial will be stopped for evaluation and consideration of revision. If at most one DLT is observed then escalation continues to the next dose level. The cohorts will escalate by 3Gy up to 21 Gy of irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Women with a biopsy proven diagnosis of low/intermediate grade ductal carcinoma in situ or invasive ductal (or other favorable histology) carcinoma of the breast
* Breast preservation candidates (no prior breast or nodal radiotherapy, no imaging evidence of multicentric or multifocal disease, no pregnant women, and no comorbid conditions precluding surgery)
* Clinical T1N0M0
* 55 years of age or older
* Estrogen receptor (ER) positive,
* No evidence of lymphovascular space invasion on initial biopsy
* Not pregnant. If not post-menopausal must adhere to birth control measures
* White blood cell count > 3000, Hemoglobin > 9, platelets >100000
* Must be eligible for MRI on initial evaluation and GFR at least 60 ml/min

Exclusion Criteria:

* Neoadjuvant chemotherapy
* Breast implants
* Medical conditions that may increase risk for poor cosmetic outcome (i.e. Lupus, rheumatoid arthritis, scleroderma)
* Patients unable to receive study treatment planning secondary to body habitus or inability to lie flat on the stomach at length
* HER-2/neu positive
* Positive serum pregnancy test

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-07-28 (Actual); Primary Completion 2016-04-04 (Actual); Study Completion 2023-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Blitzblau, MD PhD, Principal Investigator — Duke University Medical Center, Dept of Radiation Oncology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Nattinger AB, Hoffmann RG, Kneusel RT, Schapira MM. Relation between appropriateness of primary therapy for early-stage breast carcinoma and increased use of breast-conserving surgery. Lancet. 2000 Sep 30;356(9236):1148-53. doi: 10.1016/S0140-6736(00)02757-4. PMID 11030294
- [Background] Hepel JT, Tokita M, MacAusland SG, Evans SB, Hiatt JR, Price LL, DiPetrillo T, Wazer DE. Toxicity of three-dimensional conformal radiotherapy for accelerated partial breast irradiation. Int J Radiat Oncol Biol Phys. 2009 Dec 1;75(5):1290-6. doi: 10.1016/j.ijrobp.2009.01.009. Epub 2009 Apr 22. PMID 19395195
- [Background] Luini A, Orecchia R, Gatti G, Intra M, Ciocca M, Galimberti V, Veronesi P, Santos GR, Gilardi D, Veronesi U. The pilot trial on intraoperative radiotherapy with electrons (ELIOT): update on the results. Breast Cancer Res Treat. 2005 Sep;93(1):55-9. doi: 10.1007/s10549-005-3782-1. PMID 16184459
- [Derived] Horton JK, Siamakpour-Reihani S, Lee CT, Zhou Y, Chen W, Geradts J, Fels DR, Hoang P, Ashcraft KA, Groth J, Kung HN, Dewhirst MW, Chi JT. FAS Death Receptor: A Breast Cancer Subtype-Specific Radiation Response Biomarker and Potential Therapeutic Target. Radiat Res. 2015 Nov;184(5):456-69. doi: 10.1667/RR14089.1. Epub 2015 Oct 21. PMID 26488758

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Dose Radiosurgery: Dose Level 1 | Single Dose Radiosurgery: Dose Level 2 | Single Dose Radiosurgery: Dose Level 3
Started | 9 | 10 | 16
Completed | 8 | 8 | 16
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose Radiosurgery: Dose Level 1 | Single Dose Radiosurgery: Dose Level 2 | Single Dose Radiosurgery: Dose Level 3 | Total
Number analyzed (Participants) | 8 | 8 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (7.0) | 65.3 (7.1) | 67.2 (7.1) | 66.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16 | 32
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 8 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 8 | 7 | 15 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: As measured by the incidence of acute toxicity and wound healing complications
Time Frame: 30 days
Population: Participants receiving all dose levels (8 at 15Gy/Dose level 1, 8 at 18Gy/Dose level 2, 16 at 21Gy/Dose level 3)
Measure: Number; unit: Gray (Gy)
Groups:
- Single Dose Radiosurgery: All Dose Levels: A single dose of radiation in 15Gy (dose level 1), 18Gy (dose level 2) or 21Gy (dose level 3) given in radiosurgery technique about 10 days before lumpectomy.
Arm/Group | Single Dose Radiosurgery: All Dose Levels
Number analyzed (Participants) | 32
Gray (Gy) | 21

2. Secondary Outcome: Cosmetic Outcome
Description: Percent of patients with excellent or good cosmetic outcome at 3 years based on physician's assessment.
  EXCELLENT is defined as: when compared to the untreated breast or the original appearance of the treated breast, there is minimal or no difference in the size or shape of the treated breast. The way the breast feels (its texture) is the same or slightly different. There may be thickening, scar tissue, or seroma within the breast but not enough to change the appearance.
  GOOD is defined as: there is mild asymmetry between the breasts, which means that there is some acceptable difference in the size or shape of the treated breast as compared to the opposite breast or the appearance of the breast before treatment. There may be some mild reddening or darkening of the breast. The thickening or scar tissue within the breast causes a mild change in its shape or size.
Time Frame: 3 years
Population: Participants with a physician's assessment available.
Measure: Number; unit: percentage of participants
Arm/Group | Single Dose Radiosurgery: Dose Level 1 | Single Dose Radiosurgery: Dose Level 2 | Single Dose Radiosurgery: Dose Level 3
Number analyzed (Participants) | 7 | 6 | 14
percentage of participants | 71 | 100 | 100

3. Secondary Outcome: Local Control
Time Frame: 3 years
Population: Data not collected.
Arm/Group | Single Dose Radiosurgery: Dose Level 1 | Single Dose Radiosurgery: Dose Level 2 | Single Dose Radiosurgery: Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

4. Other Pre Specified Outcome: Acquire Tissue
Description: Pre and post-radiotherapy for exploratory analysis of radiation response
Time Frame: Pre and post SRS radiosurgery
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Magnetic Resonance Images(MRI)
Description: Pre and post-radiotherapy for exploratory analysis of radiation response.
Time Frame: Pre and post SRS radiosurgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Single Dose Radiosurgery: Dose Level 2: A single 18 Gy dose of radiation given in radiosurgery technique about 10 days before lumpectomy.
  Radiosurgery: Single dose or radiation in 15Gy, 18Gy or 21Gy
  Note: One participant in dose level 2 was killed in an unrelated motor vehicle accident and was not considered in all-cause mortality.
Arm/Group | Single Dose Radiosurgery: Dose Level 1 | Single Dose Radiosurgery: Dose Level 2 | Single Dose Radiosurgery: Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/8 | 1/8 | 1/16
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/16
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 15/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Dose Radiosurgery: Dose Level 1 (N=8) | Single Dose Radiosurgery: Dose Level 2 (N=8) | Single Dose Radiosurgery: Dose Level 3 (N=16)
Chest pain -cardiac (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 2
Breast infection (Infections and infestations) | 0 | 2 | 0
Infections and infestations-Other (Infections and infestations) | 0 | 1 | 1
Rash pustular (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 4 | 9
Seroma (Injury, poisoning and procedural complications) | 0 | 4 | 8
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 7 | 7 | 13
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 1 | 0 | 0
Breast atrophy (Reproductive system and breast disorders) | 2 | 1 | 3
Breast pain (Reproductive system and breast disorders) | 4 | 5 | 8
Nipple deformity (Reproductive system and breast disorders) | 1 | 0 | 0
Reproductive system and breast disorders-Other (Reproductive system and breast disorders) | 2 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 3 | 4
Skin induration (Skin and subcutaneous tissue disorders) | 3 | 1 | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hematoma (Vascular disorders) | 0 | 0 | 1
Lymphedema (Vascular disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes